CLINICAL TRIAL: NCT01924624
Title: Adjuvant Therapy With Thalidomide After Curative Resection of Hepatocellular Carcinoma.: a Randomized Controlled Trial
Brief Title: Adjuvant Therapy With Thalidomide After Curative Resection of Hepatocellular Carcinoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Xiamen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FAHXMU-013
Record Dates: First submitted 2013-07-21; First posted 2013-08-16 (Estimated); Last update posted 2013-08-16 (Estimated); Status verified 2013-07

CONDITIONS: Hepatocellular Carcinoma; Recurrence
MeSH Terms: conditions — Carcinoma, Hepatocellular; Recurrence | interventions — Thalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Thalidomide (Experimental): Thalidomide 100mg per day after the radical resection HCC
  Interventions: Drug: Thalidomide
- Control (Active Comparator): No adjuvant Thalidomide treatment after curative hepatic resection
  Interventions: Drug: Thalidomide

INTERVENTIONS:
Drug: Thalidomide — Patients in the Adjuvant group were given oral Thalidomide(at a dose of 100 mg per day) continuously during the follow-up period
  Other Names: Contergan

SUMMARY:
Postoperative recurrence of hepatocellular carcinoma (HCC) is a major problem after surgical resection. To date, adjuvant chemotherapy or other adjuvant modalities have not been proven effective in preventing or delaying recurrence. The aim of this prospective randomized study was to evaluate the effectiveness of Thalidomide as a postoperative adjuvant regimen in inhibiting the recurrence of HCC

DETAILED DESCRIPTION:
A number of modalities for preventing HCC recurrence after resection have been proposed and analyzed. Both preoperative and adjuvant transcatheter arterial chemoembolization (TACE) were found to be unable to reduce the risk of postoperative recurrence significantly, or confer a survival advantage. Vitamin K (VK) is a fat-soluble vitamin that regulates clotting factor production by acting as a coenzyme for a VK dependent carboxylase that catalyzes carboxylation of glutamic acid residues into gamma-carboxyglutamic acid. The findings in vitro have indicated that VK2 has an antiproliferative effects against hepatoma cell lines, but its efficacy in suppressing HCC recurrence was not confirmed in human studies. Interferon has a variety of biologic properties, including antiviral, immunomodulatory, antiproliferative, antiangiogenic and tumoricidal effects. It is reported that interferon is effective in preventing the development of HCC recurrence after its curative treatment in HCV-related cirrhosis. However, interferon treatment also has side-effects, including flu-like symptoms, fatigue, neutropenia, thrombocytopenia, depression, bone marrow suppression, and unmasking or exacerbation of autoimmune illnesses, which lead either to treatment disruption or dose modification. Polyprenoic acid, an acyclic retinoid, reportedly is effective in prevention of second primary hepatomas, but long-term safety and efficacy data are lacking.

Thalidomide possesses immunomodulatory,anti-inflammatory, and antiangiogenic properties.It has successfully been applied for the treatment of various malignancies including HCC.To investigated whether postoperative adjuvant therapy with Thalidomide could inhibite the recurrence of HCC after radical resection,we planed to conduct this clinical trial.

ELIGIBILITY:
Inclusion Criteria:

1. 18-75 years old,male and female
2. Patients who did not receive any anti-tumor therapies prior to the surgery (including liver transplantation, TACE, local tumor ablation, chemotherapy, radiotherapy, molecular targeted therapy and other anti-tumor therapy) resection of hepatocellular carcinoma
3. Patients who underwent radical resection of HCC, and 1 month after surgery,dynamic computed tomography showed on lesion in the liver and no signs of extrahepatic metastasis
4. Sign the informed consent

Exclusion Criteria:

1. Women who were pregnant or breast-feeding
2. signs showing recurrence or metastasis one month after surgery
3. Recurrent HCC
4. Patients unable to take drug orally
5. Patients inappropriate to participate in the trial upon the investigator's judgment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2013-07; Primary Completion 2015-08 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
disease-free survival | 5 years

SECONDARY OUTCOMES:
Overall survival | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Yanmng Zhou, MD, Principal Investigator — Xiamen University
Locations (1):
- First affiliated Hospital of Xiamen University, Xiamen, Fujian, China